CLINICAL TRIAL: NCT01209338
Title: Acceptability and Feasibility of Human Papilloma Virus Vaccine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Tata Memorial Hospital, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 655
Record Dates: First submitted 2010-06-16; First posted 2010-09-27 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sensitized group (Active Comparator): One arm will be a sensitized group which would have received cancer health awareness sessions and / or screening earlier at least once in the past.
  Interventions: Behavioral: Health education
- non-sensitized group (No Intervention): The second arm will belong to an area which has never been exposed to any form of cancer awareness or screening activities thus this group is a completely non-sensitized group.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Health education — Health education about HPV infection, HPV vaccine and cervix cancer.

SUMMARY:
The overall program goal is to determine the Acceptability and Feasibility of introducing a population based Human Papilloma Virus (HPV) Vaccination programme and understanding the key individual and community factors that would determine the potential acceptability of the vaccine.

DETAILED DESCRIPTION:
The eligible participant will be chosen by door-door household visit. Each participant will be given information regarding the study and written informed consent will be obtained from them. Their participation will be entirely voluntary and no pressure or coercion will be used. Our team will help them with questions that are not well understood by them or are ambiguous for them. The questionnaire is in 2 sections. Section one will try and ascertain the mother's Knowledge, Attitude and Perception regarding cervix cancer, HPV infection and HPV Vaccination.

Section 1 will be interviewed for a period of 5-10 minutes followed by an information sheet providing details on HPV infection, its association with cervix cancer and HPV Vaccination against cervix cancer. The information sheet available will be explained to them for a period of 10-15 minutes. Our social workers will be available at all times to allay their misinterpretations. This will be followed by section 2 which will be a post intervention questionnaire comprising of questions regarding their attitude towards HPV vaccination and identifying barriers and motivators for these women towards vaccination.

The post-intervention questionnaire would be interviewed for a period of 10-15 minutes, thus a total of 25-40 minutes will be made available to every participant for the entire session. The team is expected to cover 15 women per day totaling to 300 women per month considering the monthly holidays and time lost in certain administrative issues.

Patients will be recruited for 4 months which will be followed by data entry, data analysis, formulation of results and write -up. Thus the entire study will last for eight months. The questionnaire consists of mostly close ended questions with options in the form of yes/no/do not know. Some questions which require definitive answers have been provided with plausible options. Some questions have been left open ended so as to avoid ambiguity. The questionnaire is simple, in continuity and is translated into Hindi and Marathi languages so as to meet the needs of the local population.

ELIGIBILITY:
Inclusion Criteria:

All married women bearing daughters of the age group 10-18 years and are conversant in either Marathi, Hindi or English will be included in the study.

Exclusion Criteria:

Women with no children or with daughters outside the 10-18 yrs age group have been excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To determine the Knowledge, Attitude and Practice about cervix cancer, Human Papilloma Virus (HPV). | 8 months
  1. To determine the Knowledge, Attitude and Practice about cervix cancer, Human Papilloma Virus (HPV) and HPV Vaccines amongst the target population.
  2. To promote awareness regarding cervix cancer and its screening amongst the community.
  3. To assess the feasibility and logistics of various strategies for reaching girls with HPV Vaccines.

SECONDARY OUTCOMES:
. To identify the barriers and facilitators perceived by women for vaccinating their daughters against HPV infection and cervix cancer. | 8 months
  To determine barriers and facilitators for vaccine acceptability between sensitized and non- sensitized group.

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila A Pimple, MD, Principal Investigator — Tata Memorial Hospital; Gauravi A Mishra, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India